CLINICAL TRIAL: NCT00103610
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Comparative Trial of AMD3100 Plus G-CSF Versus G-CSF Plus Placebo to Mobilize and Collect ≥ 5 * 10^6 CD34+ Cells/kg in Non-Hodgkin's Lymphoma Patients for Autologous Transplantation
Brief Title: Mobilization of Stem Cells With AMD3100 (Plerixafor) in Non-Hodgkin's Lymphoma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMD3100-3101; NCT00248508 (obsolete NCT alias)
Record Dates: First submitted 2005-02-11; First posted 2005-02-14 (Estimated); Results first posted 2010-09-29 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-02

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Non-Hodgkin's lymphoma; Stem cell mobilization
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Granulocyte Colony-Stimulating Factor; plerixafor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- G-CSF plus plerixafor (Experimental)
  Interventions: Drug: Granulocyte colony-stimulating factor plus plerixafor
- G-CSF plus placebo (Placebo Comparator)
  Interventions: Drug: Granulocyte colony-stimulating factor plus placebo

INTERVENTIONS:
Drug: Granulocyte colony-stimulating factor plus plerixafor — Participants underwent mobilization with granulocyte colony-stimulating factor (G-CSF) (10 µg/kg/day) for 4 days, administered by subcutaneous (SC) injection. On the evening of Day 4, participants received plerixafor (240 µg/kg), administered by SC injection. On Day 5, participants received a morning dose of G-CSF (10 µg/kg) and underwent apheresis approx. 10 to 11 hours after the dose of plerixafor (within 60 minutes of G-CSF administration). Participants continued to receive an evening dose of plerixafor followed by a morning dose of G-CSF and apheresis for up to 4 aphereses or until ≥ 5*10^6 CD34+ cells/kg were collected. Participants who participated in the rescue procedure underwent an additional daily treatment with plerixafor (240 µg/kg) and apheresis for up to 4 days.
  Other Names: AMD3100; Mozobil
  Arms: G-CSF plus plerixafor
Drug: Granulocyte colony-stimulating factor plus placebo — Participants underwent mobilization with granulocyte colony-stimulating factor (G-CSF) (10 µg/kg/day) for 4 days, administered by subcutaneous (SC) injection. On the evening of Day 4, participants received placebo, administered by SC injection. On Day 5, participants received a morning dose of G-CSF (10 µg/kg) and underwent apheresis approx. 10 to 11 hours after the dose of placebo (within 60 minutes of G-CSF administration). Participants continued to receive an evening dose of placebo followed by a morning dose of G-CSF and apheresis for up to 4 aphereses or until ≥ 5*10^6 CD34+ cells/kg were collected. Participants who participated in the rescue procedure underwent an additional daily treatment with plerixafor (240 µg/kg) and apheresis for up to 4 days.
  Arms: G-CSF plus placebo

SUMMARY:
The purpose of this study is to determine whether the combination of AMD3100 (plerixafor) and granulocyte colony-stimulating factor (G-CSF or generic name filgrastim) is better than G-CSF alone to mobilize and collect the optimal number of stem cells in non-Hodgkin's lymphoma patients for autologous transplantation.

DETAILED DESCRIPTION:
A peripheral stem cell transplant may be able to replace blood-forming cells that were destroyed by chemotherapy. Currently filgrastim (G-CSF), a colony stimulating factor, is used to cause the growth and mobilization of stem cells from bone marrow to peripheral blood, which can then be collected from the peripheral blood by a process called apheresis. Plerixafor aids in the release of the stem cells from the bone marrow into the peripheral blood, possibly allowing for a more rapid collection of a larger number of stem cells from the peripheral blood. Larger stem cell doses for transplantation correlate to faster recovery times after high dose chemotherapy followed with stem cell transplantation. This study is intended to determine whether the combination of plerixafor with filgrastim is better than filgrastim alone in helping non-Hodgkin's lymphoma patients collect at least 5 million stem cells in four or less apheresis sessions.

This study was previously posted by AnorMED, Inc. In November 2006, AnorMED, Inc. was acquired by Genzyme Corporation. Genzyme Corporation is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria (Abbreviated List):

* Non-Hodgkin's lymphoma in first or second complete or partial remission
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* White Blood Cell count (WBC) > 2.5*10^9/L
* Platelet (PLT) > 100*10^9/L

Exclusion Criteria (Abbreviated List):

* Failed previous stem cell collection
* Prior autologous or allogeneic transplant
* Brain metastases or bone marrow involvement > 20%
* Radiation to pelvis
* Abnormal electrocardiogram (ECG) with rhythm disturbance (ventricular arrhythmias) or other conduction abnormality

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2005-01; Primary Completion 2006-07 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (32):
- United States (31):
  - City of Hope Samaritan Bone Marrow Transplant Program, Phoenix, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Shands Teaching Hospital, University of Florida, Gainesville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana Blood and Marrow Transplantation Center, Beech Grove, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Kansas City Cancer Center, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Medical Center: Clarkson and University Hospitals, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] DiPersio JF, Micallef IN, Stiff PJ, Bolwell BJ, Maziarz RT, Jacobsen E, Nademanee A, McCarty J, Bridger G, Calandra G; 3101 Investigators. Phase III prospective randomized double-blind placebo-controlled trial of plerixafor plus granulocyte colony-stimulating factor compared with placebo plus granulocyte colony-stimulating factor for autologous stem-cell mobilization and transplantation for patients with non-Hodgkin's lymphoma. J Clin Oncol. 2009 Oct 1;27(28):4767-73. doi: 10.1200/JCO.2008.20.7209. Epub 2009 Aug 31. PMID 19720922
- See also: Further information on non-Hodgkin's lymphoma from the National Cancer Institute — http://www.cancer.gov/cancertopics/types/non-hodgkin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with non-Hodgkin's lymphoma (NHL) eligible for autologous hematopoietic stem cell transplant were recruited from 31 centers in the U.S. and 1 in Canada. The first participant was randomized on 18 January 2005 and the last participant's last study visit occurred on 20 December 2007. A total of 298 participants were randomized.
Groups:
- G-CSF Plus Plerixafor: Participants underwent mobilization with G-CSF for 4 days. On the evening of Day 4, participants received a dose of plerixafor. On each subsequent day, participants received a morning dose of G-CSF followed by apheresis and an evening dose of plerixafor for a maximum of 4 aphereses or until ≥ 5*10^6 CD34+ cells/kg were collected.
- G-CSF Plus Placebo: Participants underwent mobilization with G-CSF for 4 days. On the evening of Day 4, participants received a dose of placebo. On each subsequent day, participants received a morning dose of G-CSF followed by apheresis and an evening dose of placebo for a maximum of 4 aphereses or until ≥ 5*10^6 CD34+ cells/kg were collected.
Period: Overall Study
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Started | 150 | 148
Completed | 112 | 68
Not Completed | 38 | 80
Not completed — Entered Rescue Procedure | 10 | 52
Not completed — Death | 16 | 12
Not completed — Elective Withdrawal | 4 | 0
Not completed — Lost to Follow-up | 3 | 1
Not completed — Adverse Event | 2 | 2
Not completed — Other | 2 | 7
Not completed — Failed mobilization | 1 | 5
Not completed — Noncompliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo | Total
Number analyzed (Participants) | 150 | 148 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (10.9) | 57.5 (10.3) | 56.3 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 46 | 96
  Male | 100 | 102 | 202
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 136 | 140 | 276
  African-American | 6 | 1 | 7
  Asian | 2 | 2 | 4
  Hispanic/Latino | 5 | 4 | 9
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Able to Achieve Target (≥ 5*10^6 CD34+ Cells/kg) in 4 or Fewer Days of Apheresis
Description: Proportion of participants achieving a target of ≥ 5*10^6 CD34+ cells/kg in 4 or fewer days of apheresis. Central lab data were taken from Days 5 to 8 of the Treatment/Apheresis period. Each participant's value was calculated as the sum of all daily values collected over the 4 apheresis days.
Time Frame: Days 5 to 8
Population: Intent-to-Treat Population
Measure: Number; unit: proportion of participants
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Number analyzed (Participants) | 150 | 148
proportion of participants
  Proportion achieving target in ≤4 days | 0.593 | 0.196
  Proportion not achieving target in ≤4 days | 0.407 | 0.804

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with treatment emergent adverse events (AEs). The timeframe for treatment emergent AEs is defined as Day 1 (start of G-CSF Mobilization) to the day before starting chemotherapy (approximately 38 days later). AEs were reported regardless of relationship to study treatment. The investigator graded each AE using the World Health Organization (WHO) Adverse Event Grading Scale. AEs of Grade 3 were considered severe and Grade 4 were considered life-threatening.
Time Frame: up to Day 38
Population: Safety population of all participants who received at least 1 mobilization dose of G-CSF or study treatment (plerixafor or placebo). Three participants did not receive G-CSF or any study treatment and were excluded from the safety analyses.
Measure: Number; unit: participants
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Number analyzed (Participants) | 150 | 145
participants
  Adverse Events (AEs) | 146 | 138
  Related AEs | 98 | 60
  AEs Leading to early treatment termination | 3 | 3
  AEs Leading to early study termination | 2 | 4
  Grade 3 (severe) or 4 (life-threatening) AEs | 11 | 14
  SAEs | 8 | 10

3. Secondary Outcome: Proportion of Participants Able to Achieve Target (>=2*10^6 CD34+ Cells/kg) in 4 or Fewer Days of Apheresis
Description: Proportion of participants achieving a target of >=2*10^6 CD34+ Cells/kg in 4 or fewer days of apheresis. Central lab data were taken from Days 5 to 8 of the Treatment/Apheresis period. Each participant's value was calculated as the sum of all daily values collected over the 4 apheresis days.
Time Frame: up to Day 8
Population: Intent-to-treat Population
Measure: Number; unit: proportion of participants
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Number analyzed (Participants) | 150 | 148
proportion of participants
  Proportion achieving target in ≤4 days | 0.867 | 0.473
  Proportion not achieving target in ≤4 days | 0.133 | 0.527

4. Secondary Outcome: Median Number of Days of Apheresis Required to Achieve >=5*10^6 CD34+ Cells/kg
Description: The Kaplan Meier estimate of median number of days (number of days at which 50% of participants reached the threshold, accounting for censored values) in each treatment arm to collect the target number of cells (≥5*10^6 CD34+ cells/kg) for transplantation. Central laboratory values were used.
Time Frame: up to Day 8
Population: Intent-to-Treat Population.
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- G-CSF + Plerixafor: Participants underwent mobilization with G-CSF for 4 days. On the evening of Day 4, participants received a dose of plerixafor. On each subsequent day, participants received a morning dose of G-CSF followed by apheresis and an evening dose of plerixafor for a maximum of 4 aphereses or until ≥ 5*10^6 CD34+ cells/kg were collected.
Arm/Group | G-CSF + Plerixafor | G-CSF Plus Placebo
Number analyzed (Participants) | 147 | 142
Days | 3.0 [1.0 to NA] — Not enough participants reached the threshold to support estimating the upper range. | NA [NA to NA] — Not enough participants reached the threshold to estimate the values.

5. Secondary Outcome: Median Number of Days to Polymorphonuclear (PMN) Cell Engraftment
Description: The Kaplan Meier estimate of median number of days to PMN engraftment (number of days at which 50% of participants have experienced the event, accounting for censored values) was a secondary efficacy endpoint. Engraftment was defined as PMN counts ≥ 0.5*10^9/L for 3 consecutive days or ≥ 1.0*10^9/L for 1 day. Time to engraftment corresponded to the first day that the criteria were met.
Time Frame: Up to Month 13
Population: Participants who received a stem cell transplant.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Number analyzed (Participants) | 135 | 82
Days | 10.0 [10.0 to 11.0] | 10.0 [10.0 to 11.0]

6. Secondary Outcome: Median Number of Days to Platelet (PLT) Engraftment
Description: The Kaplan Meier estimate of median number of days to PLT engraftment (number of days at which 50% of participants have experienced the event, accounting for censored values) was a secondary efficacy endpoint. Engraftment was defined as ≥ 20*10^9/L without transfusion for the preceding 7 days. Time to engraftment corresponded to the first day that the criteria were met.
Time Frame: Up to Month 13
Population: Participants who received a stem cell transplant
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Number analyzed (Participants) | 135 | 82
Days | 20.0 [17.0 to 25.0] | 20.0 [18.0 to 25.0]

7. Secondary Outcome: Graft Durability at 100 Days Post Transplantation
Description: The proportion of participants maintaining a durable graft at 100 days post transplantation by at least 2 of the following criteria (without erythropoietin (EPO), G-CSF, or transfusions): (1) a platelet count >50000/µL without transfusion for at least 2 weeks, (2) hemoglobin >=10g/dL for at least 1 month, (3) and absolute neutrophil count >1000/µL for at least 1 week.
Time Frame: approximately Day 138
Population: Participants who received a stem cell transplant and were evaluable at 100 days post-transplant
Measure: Number; unit: proportion of participants
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Number analyzed (Participants) | 135 | 82
proportion of participants
  Proportion of participants with durable graft | 0.948 | 0.951
  Proportion of participants without durable graft | 0.052 | 0.049

8. Secondary Outcome: Graft Durability at 6 Months Post Transplantation
Description: The proportion of participants maintaining a durable graft at 6 months post transplantation by at least 2 of the following criteria (without erythropoietin (EPO), G-CSF, or transfusions): (1) a platelet count >50000/µL without transfusion for at least 2 weeks, (2) hemoglobin >=10g/dL for at least 1 month, (3) and absolute neutrophil count >1000/µL for at least 1 week.
Time Frame: approximately Month 7
Population: Participants who received a stem cell transplant and were evaluable at 6 months post-transplant
Measure: Number; unit: proportion of participants
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Number analyzed (Participants) | 123 | 78
proportion of participants
  Proportion of participants with a durable graft | 0.976 | 0.987
  Proportion of participants without a durable graft | 0.024 | 0.013

9. Secondary Outcome: Graft Durability at 12 Months Post Transplantation
Description: The proportion of participants maintaining a durable graft 12 months post-transplantation by at least 2 of the following criteria (without erythropoietin (EPO), G-CSF, or transfusions): (1) a platelet count >50000/µL without transfusion for at least 2 weeks, (2) hemoglobin >=10g/dL for at least 1 month, (3) and absolute neutrophil count >1000/µL for at least 1 week.
Time Frame: approximately Month 13
Population: Participants who received a stem cell transplant and were evaluable at 12 months post-transplant
Measure: Number; unit: proportion of participants
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Number analyzed (Participants) | 112 | 65
proportion of participants
  Proportion of participants with a durable graft | 0.982 | 1.0
  Proportion of participants without a durable graft | 0.018 | 0.0

ADVERSE EVENTS:
Time Frame: Treatment emergent AEs covering Day 1 (start of G-CSF Mobilization to the day before starting chemotherapy (approximately Day 38).
Description: Three participants did not receive any study treatment and were excluded from the safety analyses.
  In the event a participant experienced both a serious and a non-serious form of the same AE, they were included in the numerator of both AE tables. Each AE table includes all events, regardless of reported relationship to study treatment or grade.
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Serious Adverse Events (participants affected / at risk) | 8/150 | 10/145
Other Adverse Events (participants affected / at risk) | 145/150 | 136/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | G-CSF Plus Plerixafor (N=150) | G-CSF Plus Placebo (N=145)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Catheter bacteraemia (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — A coding error occurred in coding changes from MedDRA version 6.1 to 10.0. An infectious AE coded with the preferred term bacteraemia (MedDRA version 6.1) is now coded as metastases to skin (MedDRA version 10.0).
Convulsion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | G-CSF Plus Plerixafor (N=150) | G-CSF Plus Placebo (N=145)
Anaemia (Blood and lymphatic system disorders) | 3 | 5
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 5
Angina pectoris (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Extrasystoles (Cardiac disorders) | 2 | 0
Palpitations (Cardiac disorders) | 2 | 3
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 5 | 4
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Ventricular tachyarrhythmia (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 3
Vertigo (Ear and labyrinth disorders) | 3 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Eye swelling (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 9 | 3
Abdominal pain (Gastrointestinal disorders) | 10 | 4
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 65 | 20
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 5 | 4
Dyspepsia (Gastrointestinal disorders) | 4 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 11 | 7
Frequent bowel movements (Gastrointestinal disorders) | 5 | 6
Glossodynia (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 4 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 50 | 24
Oral mucosal blistering (Gastrointestinal disorders) | 1 | 0
Oral mucosal petechiae (Gastrointestinal disorders) | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 11 | 13
Periodontitis (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Retching (Gastrointestinal disorders) | 2 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 4 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 12 | 8
Asthenia (General disorders) | 0 | 2
Catheter related complication (General disorders) | 1 | 0
Catheter site discharge (General disorders) | 2 | 3
Catheter site erythema (General disorders) | 3 | 8
Catheter site haematoma (General disorders) | 2 | 1
Catheter site haemorrhage (General disorders) | 6 | 7
Catheter site oedema (General disorders) | 0 | 3
Catheter site pain (General disorders) | 18 | 21
Catheter site pruritus (General disorders) | 2 | 3
Catheter site rash (General disorders) | 2 | 2
Catheter site related reaction (General disorders) | 2 | 4
Chest discomfort (General disorders) | 1 | 2
Chest pain (General disorders) | 0 | 2
Chills (General disorders) | 3 | 6
Fatigue (General disorders) | 40 | 33
Feeling abnormal (General disorders) | 1 | 0
Feeling cold (General disorders) | 2 | 0
Feeling hot (General disorders) | 0 | 2
Immediate post-injection reaction (General disorders) | 0 | 1
Influenza like illness (General disorders) | 2 | 2
Injection site bruising (General disorders) | 1 | 3
Injection site discomfort (General disorders) | 1 | 0
Injection site erythema (General disorders) | 48 | 10
Injection site haematoma (General disorders) | 1 | 0
Injection site haemorrhage (General disorders) | 1 | 3
Injection site irritation (General disorders) | 7 | 0
Injection site pain (General disorders) | 3 | 4
Injection site pruritus (General disorders) | 12 | 1
Injection site rash (General disorders) | 1 | 1
Injection site reaction (General disorders) | 3 | 2
Injection site swelling (General disorders) | 2 | 0
Injection site urticaria (General disorders) | 4 | 0
Local swelling (General disorders) | 1 | 0
Localised oedema (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 3
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 16 | 18
Pain (General disorders) | 12 | 15
Peripheral coldness (General disorders) | 2 | 0
Pyrexia (General disorders) | 9 | 8
Sensation of pressure (General disorders) | 1 | 0
Submandibular mass (General disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Body tinea (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Candidiasis (Infections and infestations) | 1 | 0
Catheter bacteraemia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Central line infection (Infections and infestations) | 3 | 1
Erythema induratum (Infections and infestations) | 1 | 1
Folliculitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 3
Oral candidiasis (Infections and infestations) | 1 | 1
Oral herpes (Infections and infestations) | 0 | 1
Periodontal infection (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Urinary tract infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Citrate toxicity (Injury, poisoning and procedural complications) | 3 | 2
Contusion (Injury, poisoning and procedural complications) | 5 | 4
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 3
Blood creatinine increased (Investigations) | 1 | 0
Blood magnesium decreased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
Blood pressure decreased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 2 | 8
Body temperature increased (Investigations) | 0 | 2
Breath sounds abnormal (Investigations) | 2 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 3
Urine analysis abnormal (Investigations) | 1 | 0
Weight increased (Investigations) | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 25 | 20
Hypomagnesaemia (Metabolism and nutrition disorders) | 17 | 12
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 31 | 30
Bone pain (Musculoskeletal and connective tissue disorders) | 40 | 41
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 6
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 10
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1
Areflexia (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 13 | 8
Dizziness postural (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 37 | 27
Hypoaesthesia (Nervous system disorders) | 3 | 6
Hypogeusia (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Nystagmus (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 27 | 30
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Poor quality sleep (Nervous system disorders) | 0 | 1
Sedation (Nervous system disorders) | 1 | 0
Sensory disturbance (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Syncope vasovagal (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 2 | 6
Abnormal dreams (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 7 | 7
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 2 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 11 | 4
Nightmare (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 3 | 2
Haematuria (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 1
Urine odour abnormal (Renal and urinary disorders) | 1 | 0
Breast swelling (Reproductive system and breast disorders) | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 5 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 8 | 3
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 10 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 6 | 8
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria localised (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 8 | 5
Haematoma (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 3 | 2
Hypertension (Vascular disorders) | 1 | 3
Hypotension (Vascular disorders) | 8 | 2
Pallor (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.